CLINICAL TRIAL: NCT00857233
Title: An Open-label Extension Study Examining the Safety and Tolerability of Memantine in Patients With Moderate to Severe Dementia of the Alzheimer's Type Having Completed Study 10158
Brief Title: Safety and Tolerability of Memantine in Moderate to Severe Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see explanation in the Detailed Description field.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10252
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — 20 mg oral tablets once daily
  Other Names: Ebixa®

SUMMARY:
The primary objective of the study was to examine the safety and tolerability of memantine in outpatients with moderate to severe Alzheimer's Disease.

DETAILED DESCRIPTION:
Memantine is a moderate affinity, uncompetitive N-methyl-D-aspartate (NMDA) receptor antagonist. Pre-clinical studies have demonstrated that memantine can decrease the neuronal toxicity associated with excessive glutamate release and calcium overload in neurons. Results from clinical trials in patients with moderate to severe Alzheimer's Disease (AD) have demonstrated memantine's efficacy and safety by showing positive treatment effects on cognitive, global and functional decline.

The purpose of this 24-week open-label extension study was to collect additional long-term safety and tolerability data on memantine in patients who completed the lead-in double-blind placebo-controlled Study 10158.

In agreement with Health Canada the study was prematurely terminated due to recruitment difficulties in the lead-in Study 10158. Patients ongoing in the study when the decision to terminate was taken were allowed to complete it.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory outpatients with moderate to severe dementia of the Alzheimer's type who have completed the 24-week Study 10158 and who have a knowledgeable and reliable caregiver who will accompany the patient to all clinic visits during the course of the study.

Exclusion Criteria:

* Diseases/medication which judged by the investigator could interfere with the assessments of safety, tolerability or efficacy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2004-06; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (33):
- Canada (33):
  - CA019, Edmonton, Alberta
  - CA033, Kelowna, British Columbia
  - CA043, Kelowna, British Columbia
  - CA042, Penticton, British Columbia
  - CA034, Winnipeg, Manitoba
  - CA022, Saint John, New Brunswick
  - CA045, Pictou, Nova Scotia
  - CA032, Burlington, Ontario
  - CA029, Orangeville, Ontario
  - CA004, Ottawa, Ontario
  - CA038, Peterborough, Ontario
  - CA009, Toronto, Ontario
  - CA005, Beauport, Quebec
  - CA023, Greenfield Park, Quebec
  - CA013, Montreal, Quebec
  - CA012, Sherbrooke, Quebec
  - CA030, Vanier, Quebec
  - CA017, Verdun, Quebec
  - CA015, Regina, Saskatchewan
  - CA040, Saskatoon, Saskatchewan
  - CA044, Chatham
  - CA007, Kentville
  - CA046, Kentville
  - CA001, Kingston
  - CA003, London
  - CA002, London
  - CA016, Moncton
  - CA024, Montreal
  - CA014, Montreal
  - CA011, Montreal
  - CA031, Sherbrooke
  - CA006, Toronto
  - CA037, Windsor

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an interventional, multi-centre, open-label, fixed-dose extension study to Study 10158. The Baseline visit in Study 10252 was scheduled to occur at the same time as the Week 24 Visit in Study 10158.
Pre-assignment Details: Placebo patients from Study 10158 were uptitrated in weekly increments of 5 mg over a 4-week, double-blind period. Target dose of 20 mg/day was reached at the start of the 4th week and maintained for the rest of the study. Memantine patients in Study 10158 continued on 20 mg/day. From the end of Week 4, the study was open-label.
Period: Overall Study
Arm/Group | Memantine
Started | 297
Completed | 242
Not Completed | 55
Not completed — Adverse Event | 24
Not completed — Lack of Efficacy | 1
Not completed — Non-compliance | 1
Not completed — Withdrawal of Consent | 9
Not completed — Lost to Follow-up | 4
Not completed — Nursing Home Placement | 14
Not completed — Other Reasons | 2

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 297
Age Continuous [Mean (Standard Deviation); unit: years] | 75 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 125
NPI: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Neuropsychiatric Inventory (NPI) is a validated scale that assesses behavioural disturbances in patients with dementia. The 12 item version consists of 10 behavioural and 2 neurovegetative areas. It provides both a total score as well as scores for a number of sub-scales. The frequency, severity and caregiver distress for each domain are measured. The NPI is based upon responses obtained from the caregiver. The total score is from 0 to 144. A higher score reflects more frequency and severity of the disturbances.
  Scores on a scale | 22.32 (15.41)
SIB: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a Scale] — The Severe Impairment Battery (SIB) is a validated scale used to assess cognitive function in patients with moderate to severe dementia. Items are single words or one-step commands combined with gestures. Nine domains are assessed, and the total score is between 0 and 100. A lower total score reflects the loss of cognitive function.
  Scores on a Scale | 79.99 (16.36)
CIBIC-plus: Baseline Severity Score [Mean (Standard Deviation); unit: Scores on a scale] — Clinician's Interview-Based Impression of Change-Plus Version (CIBIC-plus) is a global rating that is derived through an independent, comprehensive interview with the patient and caregiver by a rater who is barred from knowledge of all other psychometric test scores conducted as part of this protocol as well as from reported safety data. The rating is made on a 7-point scale ranging from "1 = marked improvement" to "7 = marked worsening". A score of "4" indicates no change.
  Scores on a scale | 4.52 (0.85)
ADCS-ADL - 19 items: Baseline Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) 19-item version total score for moderate to severe AD will measure patient's functioning. This battery of ADL questions is used here to measure the functional capabilities of patients with dementia. The inventory is done by interviewing a person in close contact with the patient and covers the most usual and consistent performance of the patient over the preceding 4 weeks. Total score is from 0 to 54. The higher score, the lower impairment.
  Scores on a scale | 33.43 (10.06)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: Overview of AEs
Time Frame: Baseline to Week 24
Population: Completers from lead-in study 10158 were eligible for this open-label extension study. We analysed the All-patients-treated Set (APTS) - all patients who took at least one dose of investigational medicinal product (IMP)
Measure: Number; unit: participants
Arm/Group | Memantine
Number analyzed (Participants) | 297
participants
  Patients with AEs | 191
  Patients with serious AEs (SAEs) | 27
  Patients with AEs Leading to Withdrawal | 24
  Patients with Baseline Events | 1

2. Secondary Outcome: Long-term Efficacy of Memantine on Behavioural Symptoms Using the Neuropsychiatric Inventory (NPI) - 12 Items Version Total Score.
Description: Change from Baseline in the NPI total score. Analysed by descriptive methods only.
  NPI is a validated scale that assesses behavioural disturbances in patients with dementia. The 12 item version consists of 10 behavioural and 2 neurovegetative areas. It provides both a total score as well as scores for a number of sub-scales. The frequency, severity and caregiver distress for each domain are measured. The NPI is based upon responses obtained from the caregiver. The total score is from 0 to 144. A higher score reflects more frequency and severity of the disturbances.
Time Frame: Baseline and Week 24
Population: APTS; Observed cases (OC)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 247
Scores on a scale | 2.11 (16.12)

3. Secondary Outcome: Long-term Efficacy of Memantine on Cognition Using the Severe Impairment Battery (SIB) Total Score.
Description: Change from Baseline in the SIB total score. Analysed by descriptive methods only.
  SIB is a validated scale used to assess cognitive function in patients with moderate to severe dementia. Items are single words or one-step commands combined with gestures. Nine domains are assessed, and the total score is between 0 and 100. A lower total score reflects the loss of cognitive function.
Time Frame: Baseline and Week 24
Population: APTS; OC
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 244
Scores on a scale | -5.60 (9.81)

4. Secondary Outcome: Long-term Efficacy of Memantine on Global Condition Using the Clinician's Interview-Based Impression of Change-Plus Version (CIBIC-plus).
Description: CIBIC-plus. Improvement evaluated with reference to Baseline. Analysed by descriptive methods only.
  CIBIC-plus is a global rating that is derived through an independent, comprehensive interview with the patient and caregiver by a rater who is barred from knowledge of all other psychometric test scores conducted as part of this protocol as well as from reported safety data. The rating is made on a 7-point scale ranging from "1 = marked improvement" to "7 = marked worsening". A score of "4" indicates no change.
Time Frame: Week 24
Population: APTS; OC
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 243
Scores on a scale | 4.75 (1.14)

5. Secondary Outcome: Long-term Efficacy of Memantine on Functioning Using the Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL) 19-item Version Total Score
Description: Change from Baseline on the ADCS-ADL 19-item version total score. Analysed by descriptive methods only.
  ADCS-ADL- 19 items version for moderate to severe AD will measure patient's functioning. This battery of ADL questions is used here to measure the functional capabilities of patients with dementia. The inventory is done by interviewing a person in close contact with the patient and covers the most usual and consistent performance of the patient over the preceding 4 weeks. Total score is from 0 to 54. The higher score, the lower impairment.
Time Frame: Baseline and Week 24
Population: APTS; OC
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 247
Scores on a scale | -4.16 (6.45)

6. Primary Outcome: Percentage of Patients Who Withdrew Due to Intolerance to Treatment
Time Frame: Baseline to Week 24
Population: APTS
Measure: Number; unit: percentage of participants
Arm/Group | Memantine
Number analyzed (Participants) | 297
percentage of participants | 8.1

ADVERSE EVENTS:
Time Frame: 24 weeks plus 30 days safety follow-up period
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 27/297
Other Adverse Events (participants affected / at risk) | 85/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=297)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Hip fracture (Injury, poisoning and procedural complications) | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dementia Alzheimer's type (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Social stay hospitalisation (Social circumstances) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=297)
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 10
Gait disturbance (General disorders) | 9
Fall (Injury, poisoning and procedural complications) | 15
Dizziness (Nervous system disorders) | 15
Headache (Nervous system disorders) | 10
Agitation (Psychiatric disorders) | 18
Confusional state (Psychiatric disorders) | 10

LIMITATIONS AND CAVEATS:
Long recruitment, premature termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications. Order of authors has to be established. Publication of the results by the investigator will be subject to mutual agreement between the investigator and H. Lundbeck A/S. Manuscripts and abstracts must be sent to H. Lundbeck A/S at least one month prior to submission for publication or presentation.